CLINICAL TRIAL: NCT03145090
Title: Interest of Bone Scintigraphy in Pre-operative Assessment of Knee Osteoarthritis in Patients Undergoing Unicompartmental Knee Arthroplasty
Brief Title: Bone Scintigraphy and Unicompartimental Knee Arthroplasty
Acronym: PUC-INTEVO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PUC-INTEVO (29BRC17.0027)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2018-07

CONDITIONS: Bone Scintigraphy and Knee Arthroplasty
Keywords: bone scintigraphy; knee arthroplasty; spect-ct; quantification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study the potential interest of bone scintigraphy for patients undergoing unicompartmental knee arthroplasty

DETAILED DESCRIPTION:
Knee osteoarthritis is a very common disease with significant functional consequences. Surgical treatment is the ultimate treatment with the possibility of replacing only one compartment or the 3 joint compartments.

Consequently, the pre-surgical imaging is essential to ensure that the 3 compartments are not compromised when a uni-compartmental prosthesis (PUC) is considered.

The scintigraphy because of its good diagnostic performance seems to be interesting in this indication for the preoperative assessment of knee uni-compartmental prostheses to ensure the absence of degenerative lesion of the unoperated compartment.

This study will evaluate the impact of bone scintigraphy on surgery and the potential correlation between scintigraphic and clinical data; study the pronostic impact of bone scintigraphy

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years old / uni or bilateral unicompartmental knee prothesis/ non opposition

Exclusion Criteria:

* Under 18 years old/ contraindications for bone scintigraphy/ refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient over 18 years old undergoing unicompartmental knee arthroplasty (1 or 2 knee) and who accept the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
modification in surgical strategy according to bone scintigraphy results | 18 months
  pourcentage of therapeutic modification according to bone scintigraphy results

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - Clinique de La Baie, Morlaix